CLINICAL TRIAL: NCT02891811
Title: A Randomized Phase II, 2-armed Study in Transplant Ineligible (TI) Patients With Newly Diagnosed Multiple Myeloma (NDMM) Comparing Carfilzomib + Thalidomide + Dexamethasone (KTd) Versus Carfilzomib + Lenalidomide + Dexamethasone (KRd) Induction Therapy With Respect to Response Rates and Investigating a Carfilzomib (K) Monotherapy Maintenance Strategy
Brief Title: Patients With Newly Diagnosed Multiple Myeloma Comparing KTd vs. KRd Induction Therapy and Investigating a K-mono Maintenance Strategy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_MM-2; 2016-000475-24 (EudraCT Number)
Record Dates: First submitted 2016-08-10; First posted 2016-09-08 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma
Keywords: newly diagnosed multiple myeloma; carfilzomib; thalidomide; lenalidomide; dexamethasone; transplant ineligible; induction therapy; maintenance; Study Group of Medical Tumour Therapy (AGMT)
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Thalidomide; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction Arm A (Experimental): Carfilzomib + Thalidomide + Dexamethasone (KTd) for 9 cycles (day 1-28) Followed by second randomisation: maintenance arm with carfilzomib monotherapy versus "observation only" arm
  Interventions: Drug: Carfilzomib; Drug: Thalidomide; Drug: Dexamethasone
- Induction Arm B (Active Comparator): Carfilzomib + Lenalidomide + Dexamethasone (KRd) for 9 cycles (day 1-28) Followed by second randomisation: maintenance arm with carfilzomib monotherapy versus "observation only" arm
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Induction treatment: Cycle 1 day 1+2: 20 mg/m2; days 8,9, 15 and 16: 27 mg/m2; Cycle 2: 27 mg/m2 on days 1,2,8,9,15 and 16; Cycle 3-9: 56 mg/m2 on days 1, 8 and 15; IV duration: 30-60 minutes; Maintenance treatment with carfilzomib (last tolerated dose on day 1 and 15 (± 7 days) of each cycle)
  Other Names: Kyprolis
Drug: Thalidomide — 100mg orally on days 1-28 in patients <75 years of age at Cycle 1; 50mg p.o. on days 1-28 in patients ≥ 75 years of age at Cycle 1
  Arms: Induction Arm A
Drug: Lenalidomide — 25mg p.o. on days 1-21 of each cycle
  Arms: Induction Arm B
Drug: Dexamethasone — 40mg p.o. on days 1, 8, 15,22 (± 1 day ) in patients <75 years of age at Cycle 1; 20mg p.o. on days 1, 8, 15, 22 (± 1 day) in patients ≥ 75 years of age at Cycle 1, given 4 hours-30 min prior to carfilzomib

SUMMARY:
This is a randomized, 2-arm phase II, multi-center study to evaluate the overall response rate in newly diagnosed, transplant ineligible patients receiving 9 cycles induction therapy with either KTd or KRd followed by randomization to either carfilzomib maintenance treatment for 12 months or to observation only. Maintenance is given for 12 cycles or progression of disease, whatever occurs first.

DETAILED DESCRIPTION:
Multiple myeloma, a clonal neoplastic proliferation of plasma cells, is the second most common hematologic malignancy and accounts for approximately 72,000 annual deaths worldwide. There are an estimated 11,000 deaths per year in the US and more than 19,000 deaths per year in Europe.

This study examines the efficacy of carfilzomib (K) in combination with thalidomide, an old, well established first line immunomodulatory imide drugs (IMiD) in newly diagnosed multiple myeloma versus K in combination with lenalidomide in 1st line. This trial will also evaluate the adherence to and the safety of a thalidomide containing triplet by using a non-neurotoxic proteasome inhibitor. Moreover, weekly dosing of carfilzomib addresses the need for a more convenient dosing schedule. Finally, yet importantly, this trial will assess the efficacy of a less cost intensive triplet and a strategy to keep lenalidomide as backup for later lines.. The second part of the study - after completing 9 cycles induction therapy with KTd or KRd - patients of both arms will be pooled and again randomized 1:1 stratified by induction therapy into two arms (K-monotherapy versus observation-only).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent in accordance with federal, local, and institutional guidelines
* newly diagnosed, symptomatic multiple myeloma
* Transplant-ineligibility: age > 65 years or patients not eligible due to comorbidities determined by investigator or patients not willing to undergo autologous stem-cell transplantation (ASCT) on personal preference
* Measurable disease, as defined by one or more of the following (assessed within 21 days prior to randomization):

  * Serum M-protein ≥ 0.5 g/dL, or
  * Urine M-protein ≥ 200 mg/24 hours, or
  * In subjects without detectable serum or urine M-protein, serum-free light chain (SFLC) > 100 mg/L (involved light chain) and an abnormal κ/λ ratio
* No prior treatment for multiple myeloma
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1
* Patients at cardiac risk (NYHA >II or pre-existing coronary heart disease or any other relevant cardiac complication) should be scheduled for a baseline echocardiography (ECHO) and can only be included if the left ventricular ejection fraction (LVEF) is ≥40%); independent of cardiac risk ECG has to be done for inclusion of Asian patients and patients > 75 years of age
* Adequate organ and bone marrow function within the 21 days prior to randomization defined by:

  * Bilirubin < 2 times the upper limit of normal (ULN), Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times the ULN
  * growth factor support for max 3 days allowed to achieve an absolute neutrophil count (ANC) ≥ 1000/mm3 (screening ANC should be of required)
  * Hemoglobin ≥ 7.0 g/dL; use of erythropoietic stimulating factors and red blood cell (RBC) transfusion per institutional guidelines is allowed, however the most recent RBC transfusion may not have been done within 7 days prior to obtaining screening hemoglobin.
  * Platelet count ≥ 30,000/mm3
* Calculated or measured creatinine clearance (CrCl) of ≥ 30 mL/min. Calculation should be based on the Cockcroft and Gault formula: [(140 - Age) ∙ Mass (kg) / (72 ∙ Creatinine mg/dL)]; multiply result by 0.85 if female
* Females of childbearing potential (FCBP) must have a confirmed negative serum pregnancy test within the 21 days prior to randomization (performed at a central laboratory).
* Females of childbearing potential and male subjects who are sexually active with FCBP must agree to use effective concomitant method(s) of contraception during the study and for 30 days (women) and 90 days (men) following the last study drug treatment administration.

Exclusion Criteria:

* ECOG ≥2
* Frail patients
* Waldenström macroglobulinemia
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Plasma cell leukemia (> 2.0 × 109/L circulating plasma cells by standard differential)
* Myelodysplastic syndrome
* Smoldering myeloma and monoclonal gammopathy of undetermined significance (MGUS)
* Second malignancy within the past 5 years except:

  * Adequately treated basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Prostate cancer ≤ Gleason score 6 with stable prostate-specific antigen (PSA over 12 months
  * Ductal breast carcinoma in situ with full surgical resection (i.e., negative margins)
  * Treated medullary or papillary thyroid cancer
  * Similar condition with an expectation of > 95% five-year disease-free survival
* History of or current amyloidosis
* Immunotherapy within the 21 days prior to randomization
* Glucocorticoid therapy within the 14 days prior to randomization that exceeds accumulative dose of 160 mg dexamethasone or 1000 mg prednisone
* Extended field radio therapy (more than 3 fields) within the 21 days prior to randomization
* Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib) or any other component of formulation
* Contraindication to dexamethasone, thalidomide or lenalidomide or any of the required concomitant drugs, supportive treatments or antiviral drugs, also including contraindication or hypersensitivity to any other components of these drugs (eg. hereditary galactose intolerance, complete lactase deficiency or glucose-galactose malabsorbtion in case of excipient lactose)
* Active congestive heart failure (New York Heart Association [NYHA] Class III or IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, acute diffuse infiltrative pulmonary disease, pericardial disease, or myocardial infarction within 4 months prior to enrollment
* Active infection within the 14 days prior to randomization requiring systemic antibiotics and/or antiviral therapy
* Pleural effusions requiring thoracentesis within the 14 days prior to randomization
* Ascites requiring paracentesis within the 14 days prior to randomization
* Uncontrolled hypertension or uncontrolled diabetes despite medication
* Significant neuropathy (Grade 2 with pain or Grade 3 or higher) within the 14 days prior to randomization
* Known cirrhosis
* Known human immunodeficiency virus (HIV) seropositivity, hepatitis C infection, or hepatitis B infection: subjects with past hepatitis B virus (HBV) infection or resolved HBV infection defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen (HBc) antibody test are eligible; subjects positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Participation in another interventional study within the 28 days prior to randomization
* Major surgery (except kyphoplasty) within the 28 days prior to randomization
* Female subjects who are pregnant or lactating
* Any other clinically significant medical disease or social condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent, be compliant with study procedures, or provide accurate information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Response Rates | 36 weeks after start of induction treatment (9 cycles, each cycle is 28 days)
  Overall response rate (ORR) will be assessed according to International Myeloma Working Group (IMWG) criteria to determine the ORR in patients NDMM after receiving 9 cycles induction therapy with either carfilzomib in combination with thalidomide and dexamethasone or carfilzomib in combination with lenalidomide and dexamethasone

SECONDARY OUTCOMES:
Feasibility of a carfilzomib monotherapy maintenance | after 12 months of maintenance therapy or observation only
  Feasibility of maintenance therapy with carfilzomib will be investigated in comparison with observation only strategy by observing treatment and visit compliance (listing withdrawals, treatment/visit delays and drug modifications).
Safety (adverse events) of a carfilzomib monotherapy maintenance | after 12 months of maintenance therapy or observation only
  Safety will be assessed by the type, incidence, severity (CTCAE v 4.0), and relatedness of adverse events (AEs) to treatment and by the descriptive analysis of laboratory parameters related to safety. Adverse events will be summarized by presenting the number and percentage (as appropriate) of patients having any adverse event by body system, type of adverse event, and maximum severity.
Overall response rate (efficacy) of a carfilzomib monotherapy maintenance | after 12 months of maintenance therapy or observation only
  After 12 months maintenance treatment or observation overall response rate (ORR, ratio of the number of patients with CR to partial response (PR) divided by the number of all patients evaluable for response) will be analyzed descriptively and compared using a chi^2 test without continuity correction. A one-sided 97.5% confidence interval for the difference in ORR will be calculated.
Response | after 21 months (9 months induction therapy and 12 months maintenance)
  The updated IMWG response criteria will be applied for response evaluation in all patients; this also includes minimal residual disease (MRD) evaluation; thus, response rates will be assessed qualitatively and quantitatively; MRD testing will be performed in all patients achieving complete remission (CR) and in patients which are in a CR at the end of maintenance
Overall survival (OS) | after 21 months (9 months induction therapy and 12 months maintenance)
  To determine Overall Survival (OS) in patients with NDMM ineligible for transplantation receiving either KTd versus KRd induction therapy and sub-sequent being randomised either to maintenance arm with carfilzomib or to control only for a maximum period of 12 months.
Progression free survival (PFS) | after 9 months induction therapy
  Response rates will be assessed qualitatively and quantitatively (PR, VGPR, CR, sCR, MRD according to IMWG Rajkumar 2011)
Safety and tolerability (adverse events) of induction and maintenance treatment | after 21 months (9 months induction therapy and 12 months maintenance)
  Safety and tolerability of KTd and KRd followed by randomization to carfilzomib maintenance for a maximum period of 12 months or observation only will be assessed by the type, incidence, severity (CTCAE v 4.0), and relatedness of AEs to treatment and by the descriptive analysis of laboratory parameters related to safety. Adverse events will be summarized by presenting the number and percentage (as appropriate) of patients having any adverse event by body system, type of adverse event, and maximum severity.
Changes in quality of life (QoL) | after 21 months (9 months induction therapy and 12 months maintenance)
  Changes in quality of life will be analyzed by using the cancer patient-specific questionnaire EORTC-QLQ-C30. Measures will be calculated and analyzed descriptively, and compared between treatment groups using a Mann-Whitney U-test for unpaired observations.
Changes in quality of life (QoL) using multiple myeloma specific questionnaire | after 21 months (9 months induction therapy and 12 months maintenance)
  Changes in quality of life will be analyzed by using the multiple myeloma-specific questionnaire "EORTC-QLQ-MY20". Measures will be calculated and analyzed descriptively, and compared between treatment groups using a Mann-Whitney U-test for unpaired observations.
Changes of general health status | after 21 months (9 months induction therapy and 12 months maintenance)
  Changes in general health status will be analyzed by using the questionnaires "EQ-5D-5L". QoL measures will be calculated and analyzed descriptively, and compared between treatment groups using a Mann-Whitney U-test for unpaired observations.

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Ludwig, MD, Study Director — Wilhelminenspital Vienna
Locations (21):
- Austria (19):
  - Medizinische Universitaet Graz, Univ.-Klinik f. Innere Medizin, Onkologie, Graz
  - Med. Universität Innsbruck, Univ.-Klinik f. Innere Medizin V, Hämatologie u. Onkologie, Innsbruck
  - Bezirkskrankenhaus Kufstein, Innere Medizin, Interne II u. onkologische Tagesklinik, Kufstein
  - LKH Hochsteiermark - Standort Leoben Abteilung für Innere Medizin und Hämatologie und internistische Onkologie, Leoben
  - Ordensklinikum Linz - Barmherzige Schwestern Linz, Interne I, Linz
  - Ordensklinikum Linz - Elisabethinen, I. Interne Abt. Haemato-Onkologie, Linz
  - Kepler Univ.-Klinikum Linz, Klinik f. Interne 3, Linz
  - Univ.Klinikum Krems, Klin. Abt. f. Innere Medizin 2, Mitterweng
  - Landeskrankenhaus Rankweil, Interne E (Hämatologie u. Onkologie), Rankweil
  - PMU Salzburg, Salzburg
  - Univ.-Klinikum St. Pölten, Innere Medizin 1, Sankt Pölten
  - Pyhrn-Eisenwurzen Klinikum Steyr, Innere Medizin II Onkologie, Steyr
  - Medizinische Univ. Wien, Univ.Klinik f. Innere Medizin I, Onkologie, Vienna
  - Hanusch-Krankenhaus, Vienna
  - Sozialmedizinisches Zentrum Ost - Donauspital, 2. Medizinische Abteilung, Vienna
  - Medizinische Univ. Wien, Univ.Klinik f. Innere Medizin I, Hämatologie u. Hämostaseologie, Vienna
  - Wilhelminenspital, Vienna
  - Landesklinikum Wiener Neustadt, Abteilung Onkologie, Wiener Neustadt
  - Krankenhaus Zams, Innere Medizin, Internistische Onkologie u. Hämatologie, Zams
- Germany (2):
  - UK Leipzig Medizinische Klinik und Poliklinik I, Leipzig
  - UK Würzburg Medizinische Klinik und Poliklinik II, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor — http://www.agmt.at